CLINICAL TRIAL: NCT04840823
Title: A Randomized, Double-blind, Parallel Group, Single Centre, Phase 1b/2 Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Three Orally Administered Doses of Enoxacin (200mg Twice Daily, 400mg Twice Daily and 600mg Twice Daily) in Adults With Amyotrophic Lateral Sclerosis
Brief Title: Enoxacin for Amyotrophic Lateral Sclerosis (ALS)
Acronym: REALS-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Weizmann Institute of Science (Other); Apotex Inc. (Industry)
Responsible Party: Principal Investigator, Angela Genge, Associate Professor, Neurologist, Neurology and Neurosurgery, McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REALS-1
Record Dates: First submitted 2021-03-29; First posted 2021-04-12 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Enoxacin
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Enoxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enoxacin 200mg twice daily (Experimental): Enoxacin 200mg twice daily (one dose in the morning and one dose in the evening) for 30 days, except day 1 and day 30 when only the morning dose will be taken. Participants will take 1 active 200mg enoxacin tablet and 2 placebo tablets per dose.
  Interventions: Drug: Enoxacin; Drug: Placebo
- Enoxacin 400mg twice daily (Experimental): Enoxacin 400mg twice daily (one dose in the morning and one dose in the evening) for 30 days, except day 1 and day 30 when only the morning dose will be taken. Participants will take 2 active 200mg enoxacin tablets and 1 placebo tablet per dose.
  Interventions: Drug: Enoxacin; Drug: Placebo
- Enoxacin 600mg twice daily (Experimental): Enoxacin 600mg twice daily (one dose in the morning and one dose in the evening) for 30 days, except day 1 and day 30 when only the morning dose will be taken. Participants will take 3 active 200mg enoxacin tablets per dose.
  Interventions: Drug: Enoxacin

INTERVENTIONS:
Drug: Enoxacin — Oral 200mg tablet
Drug: Placebo — Oral tablet
  Arms: Enoxacin 200mg twice daily; Enoxacin 400mg twice daily

SUMMARY:
The study will assess the safety of the drug enoxacin at specific dose levels in adults with ALS.

DETAILED DESCRIPTION:
Participants will be randomized to one of three doses of enoxacin (200, 400, or 600mg twice daily) for 30 days. On day 1, 7, 14, 21, and 30 of treatment and at a follow-up visit 14 days after the last dose, participants will be assessed for safety measures and blood will be collected to assist with the determination of enoxacin pharmacokinetics (PK) and pharmacodynamics (PD). On day 1 and day 30 of dosing, participants will only take one dose of study medication (the morning dose) to assist with determination of enoxacin single dose PK over a 24-hour period. A lumbar puncture (LP) to collect cerebrospinal fluid (CSF) for PD assessments will occur on day 1 and day 30.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of familial or sporadic ALS
* FVC of ≥ 50 percent predicted
* If female, is not breastfeeding and is not pregnant
* Has been on a stable dose of riluzole, or has not taken riluzole, for at least 30 days prior to screening
* If taking concomitant edaravone at study entry, must have completed at least one cycle of edaravone therapy prior to screening
* Not currently taking and has not taken for at least 30 days prior to screening any Theophylline containing medications, clozapine, or duloxetine
* No active infection in the 30 days prior to randomization
* Has not taken any fluoroquinolone antibiotics for at least 30 days prior to screening

Exclusion Criteria:

* Hypersensitivity/allergy to fluoroquinolones
* Diagnosed with another neurodegenerative disease
* Significant pulmonary disorder not attributed to ALS, central nervous system disorder associated with seizures, myasthenia gravis, active rheumatologic disease, tendinopathy, or any severe uncontrolled medical condition (other than ALS)
* Severe renal impairment or impaired liver function
* Baseline prolongation of QT interval/corrected QT interval (QTc) at screening, treatment with any agent that may prolong Qt/QTc interval, or history of any other at-risk other cardiac condition
* Currently enrolled in another clinical trial involving an experimental drug or device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | From baseline (prior to dosing on day 1 of dosing) to 14 day +/- 2 day follow up visit
  The incidence of adverse events (new or worsened from baseline (where baseline refers to those AEs recorded prior to dosing on day 1 of dosing)) will be summarized by primary system organ class and preferred term as frequency count and percentage of participants with AEs.
Incidence of abnormalities in clinical laboratory assessments | From baseline (prior to dosing on day 1 of dosing) to 14 day +/- 2 day follow up visit
  Clinical laboratory data will be characterized by abnormalities in values and in changes from baseline values, where baseline refers to measurements taken prior to dosing on day 1 of dosing.
Incidence of abnormalities in vital signs | From baseline (prior to dosing on day 1 of dosing) to 14 day +/- 2 day follow up visit
  Vital sign data will be characterized by abnormalities in values and in changes from baseline values, where baseline refers to measurements taken prior to dosing on day 1 of dosing.
Incidence of abnormalities in physical and neurological examinations | From baseline (prior to dosing on day 1 of dosing) to 14 day +/- 2 day follow up visit
  Physical and neurological examinations will be characterized by abnormalities and in changes from baseline, where baseline refers to measurements taken prior to dosing on day 1 of dosing.
Incidence of abnormalities in electrocardiograms (ECGs) | From baseline (prior to dosing on day 1 of dosing) to 14 day +/- 2 day follow up visit
  ECG data will be characterized by abnormalities in values and in changes from baseline values, where baseline refers to measurements taken prior to dosing on day 1 of dosing.
Ability of participants to remain on their assigned dose for the full 30 day treatment period | From the beginning (day 1) to the end (day 30) of the 30 day treatment period
  The ability of participants to remain on each dose level will be measured by the mean number of missed doses.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of enoxacin after administration on day 1 and 30 | Prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing.
  Enoxacin plasma concentrations measured in each individual participant prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing will be used to derive the Cmax.
Time of maximum plasma concentration (Tmax) of enoxacin after administration on day 1 and 30 | Prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing.
  Enoxacin plasma concentrations measured in each individual participant prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing will be used to derive the Tmax.
Area under the plasma concentration-time curve from time zero until the time corresponding with the last observed quantifiable concentration (AUC 0-last) of enoxacin after administration on day 1 and 30 | Prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing.
  Enoxacin plasma concentrations measured in each individual participant prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing will be used to derive the (AUC) 0-last.
Area under the plasma concentration-time curve extrapolated to infinity (AUC 0-inf) of enoxacin after administration on day 1 and 30 | Prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing.
  Enoxacin plasma concentrations measured in each individual participant prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing will be used to derive the AUC 0-inf.
Terminal half-life (t1/2) of enoxacin after administration on day 1 and 30 | Prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing.
  Enoxacin plasma concentrations measured in each individual participant prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing will be used to derive the t1/2.
Accumulation ratio (R) of enoxacin after administration on day 1 and 30 | Prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing.
  Enoxacin plasma concentrations measured in each individual participant prior to dosing and at 1, 2, 4, 6, 8 and 24 hours post morning dosing on days 1 and 30 of dosing will be used to derive the R.
Trough plasma concentration at pre-dose of enoxacin on day 7, 14, 21, and 30 | Prior to morning dosing on days 7, 14, 21, and 30.
  Enoxacin plasma concentrations measured in each individual participant prior to morning dosing on days 7, 14, 21, and 30 will be used to derive the trough plasma concentration at pre-dose.
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) score at baseline and at the end of the follow-up period | At baseline (prior to dosing on day 1 of dosing) and at the 14 day +/- 2 day follow-up visit
  The ALSFRS-R will be used to measure activities of daily living (ADL) and global function across four domains (respiratory, bulbar function, gross motor skills, and fine motor skills) and consists of 12 questions, each scored from 0 to 4, for a total possible score of 48, with higher scores representing better function.
King's College (KINGS) stage at baseline and at the end of the follow-up period | At baseline (prior to dosing on day 1 of dosing) and at the 14 day +/- 2 day follow-up visit
  The KINGS staging system for ALS will be used to assess the course of the disease and is based on the number of involved regions (where the three possible regions are bulbar, upper limb or lower limb) for the first three stages and the need for gastrostomy and non-invasive ventilation for the subsequent stages. The possible stages in the KINGS staging system are as follows: Stage 1: First Region Involved; Stage 2: Second Region Involved; Stage 3: Third Region Involved; Stage 4a: Nutritional Failure (need for gastrostomy); Stage 4b: Respiratory Failure (need for non-invasive ventilation); and Stage 5: Death.
Forced Vital Capacity (FVC) measurements at baseline and at the end of the follow-up period | At baseline (prior to dosing on day 1 of dosing) and at the 14 day +/- 2 day follow-up visit

OTHER OUTCOMES:
Ability of enoxacin to modulate the expression of one or more miRNA species in cerebrospinal fluid (CSF) and/or plasma | Blood: prior to morning dosing on days 1, 7 (+/- 2 days), 14 (+/- 2 days), 21 (+/- 2 days) and 30, and at the 14 day +/- 2 day follow-up visit. CSF: prior to dosing on day 1, and 2 hours (+/-1 hour) post dosing on day 30.
  Expression levels of miRNA species will be measured in CSF and/or plasma

CONTACTS AND LOCATIONS:
Overall Officials: Angela Genge, MD, FRCP, Principal Investigator — McGill University
Locations (1):
- Montreal Neurological Institute-Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haramati S, Chapnik E, Sztainberg Y, Eilam R, Zwang R, Gershoni N, McGlinn E, Heiser PW, Wills AM, Wirguin I, Rubin LL, Misawa H, Tabin CJ, Brown R Jr, Chen A, Hornstein E. miRNA malfunction causes spinal motor neuron disease. Proc Natl Acad Sci U S A. 2010 Jul 20;107(29):13111-6. doi: 10.1073/pnas.1006151107. Epub 2010 Jun 29. PMID 20616011
- [Background] Emde A, Eitan C, Liou LL, Libby RT, Rivkin N, Magen I, Reichenstein I, Oppenheim H, Eilam R, Silvestroni A, Alajajian B, Ben-Dov IZ, Aebischer J, Savidor A, Levin Y, Sons R, Hammond SM, Ravits JM, Moller T, Hornstein E. Dysregulated miRNA biogenesis downstream of cellular stress and ALS-causing mutations: a new mechanism for ALS. EMBO J. 2015 Nov 3;34(21):2633-51. doi: 10.15252/embj.201490493. Epub 2015 Sep 1. PMID 26330466
- [Background] Reichenstein I, Eitan C, Diaz-Garcia S, Haim G, Magen I, Siany A, Hoye ML, Rivkin N, Olender T, Toth B, Ravid R, Mandelbaum AD, Yanowski E, Liang J, Rymer JK, Levy R, Beck G, Ainbinder E, Farhan SMK, Lennox KA, Bode NM, Behlke MA, Moller T, Saxena S, Moreno CAM, Costaguta G, van Eijk KR, Phatnani H, Al-Chalabi A, Basak AN, van den Berg LH, Hardiman O, Landers JE, Mora JS, Morrison KE, Shaw PJ, Veldink JH, Pfaff SL, Yizhar O, Gross C, Brown RH Jr, Ravits JM, Harms MB, Miller TM, Hornstein E. Human genetics and neuropathology suggest a link between miR-218 and amyotrophic lateral sclerosis pathophysiology. Sci Transl Med. 2019 Dec 18;11(523):eaav5264. doi: 10.1126/scitranslmed.aav5264. PMID 31852800
- See also: Clinical Research Unit at The Montreal Neurological Institute-Hospital, McGill University — https://cru.mcgill.ca/